CLINICAL TRIAL: NCT02885818
Title: Does Abatacept Induce Regulatory B Cells in Patients With Rheumatoid Arthritis
Acronym: ABATACEPT_B
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ABATACEPT AND B CELL
Record Dates: First submitted 2016-08-22; First posted 2016-09-01 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Abatacept disrupts T-cell coactivation signals in rheumatoid arthritis (RA). Its potential effects on B cells are not well described. This study will assess the effects of abatacept therapy on the phenotype and function of peripheral blood B cells in patients with RA.

ELIGIBILITY:
Inclusion Criteria:

* RA as defined by ACR/EULAR criteria
* Clinical indication to start abatacept therapy

Exclusion Criteria:

* Treatment by rituximab in the previous year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA fulfilling ACR/EULAR criteria, in whom abatacept is started as part of their usual clinical care
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Peripheral blood B-cell phenotype changes | 3 months
  Measure of the proportion of the main B-cell subsets (transitional, naïve, memory, plasmablasts) by FACS analysis before abatacept initiation and 3 months later.

SECONDARY OUTCOMES:
In vitro B-cell function and regulatory properties | 3 months
  In vitro culture of B cells from the patients to assess B cell inhibition of T cell proliferation before abatacept initiation and 3 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques-Olivier Pers, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No